CLINICAL TRIAL: NCT03843281
Title: Efficacy of Paracetamol in Addition to Morphine to Improve Analgesia in the Emergency Department: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Paracetamol in Addition to Morphine to Improve Analgesia in the Emergency Department
Acronym: ParaMoED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bruno Minotti (Other)
Responsible Party: Sponsor-Investigator, Bruno Minotti, Sponsor-Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTU17.014
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Analgesia
Keywords: Paracetamol; Morphine
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Sodium Chloride; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol 1 g (100 mL) IV + Morphine 0.1 mg/kg IV (repeatable in Doses of 0.05 mg/kg), 100 patients over 4 hours
  Interventions: Drug: Paracetamol; Drug: Morphine
- Placebo (Placebo Comparator): Placebo (NaCl 0.9% 100 mL IV) + Morphine 0.1 mg/kg IV (repeatable in Doses of 0.05 mg/kg), 100 patients over 4 hours
  Interventions: Drug: Placebo; Drug: Morphine

INTERVENTIONS:
Drug: Paracetamol — s. above
  Other Names: Paracetamol Sintetica
  Arms: Paracetamol
Drug: Placebo — s. above
  Other Names: NaCl 0.9%
  Arms: Placebo
Drug: Morphine — s. above
  Other Names: Morphine Sintetica

SUMMARY:
The purpose of this study is to test the additional effect of paracetamol in combination with morphine for analgesia, respectively to test/confirm an opioid sparing effect due to the additional use of Paracetamol, as well as the reduction of adverse drug reactions of morphine.

DETAILED DESCRIPTION:
Paracetamol (acetaminophen) is widely used around the world for mild to moderate pain in all age groups. Prescription at the emergency department is very common and some studies suggest the use in alternative of Morphine, at least in the renal colic.

Morphine has also a complex analgesic effect due to inhibition of µ Receptors in the central nervous system and in the dorsal horn of the spinal cord. Morphine (like other opioids) is accepted as a cornerstone of acute pain management in the emergency department. However, occurrence of adverse drug reactions is up to 25%, mainly nausea and drowsiness.

The use of paracetamol in addition to morphine showed in a meta-analysis in the post-operative setting an opioid sparing effect of 20% over the first postoperative 24 hours, but did not change the incidence of morphine-related adverse effects in the postoperative period. An additive effect was showed of the two medicaments in another Study measuring the median effective analgesic dose (ED50).

The purpose of this study is to test the additional effect of paracetamol in combination with morphine for analgesia, respectively to test/confirm an opioid sparing effect due to the additional use of Paracetamol, as well as the to reduction of adverse drug reactions of morphine.

The study is a multicenter, randomized, double-blind, placebo-controlled. We randomize patients with pain-score >=4 on a pain Scala of 0-10 Points (numeric rating scale) in two group, one with paracetamol, one with placebo to investigate the (additive) effect of paracetamol in combination with morphine. The treatment team and the patients will be blinded to the administration. The study design is outlined to confirm the result of previous studies who stated a 20% reduction of morphine doses when combined with paracetamol. Study duration for each patient would be 240 min.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pain with Pain-score is more or equal than four in a numeric rating scale from zero to ten (i.e. indication for a treatment with morphine)
* Age over 18
* Signed informed consent. In case, patient is not able to sign the informed consent due to pain, at least verbal consent has to be provided. After pain relief, written informed consent with data and time has to be obtained

Exclusion Criteria:

* Analgesia in the past last 6 hours prior to visit at the emergency department
* Current Analgesia with long-acting/extended-release drugs
* Current Analgesia with opioids
* Chronic pain syndrome
* Contraindication for either paracetamol or morphine
* Patient's refusal of paracetamol or morphine treatment
* Pregnancy or Breastfeeding
* GCS < 13
* SpO2 < 90% with a maximum of 4 L/Min O2
* Systolic Blood Pressure < 90 mmHg
* "Fast Track"/Notfallpraxis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the total dose of morphine till pain < 4 on the NRS (0-10) after the first infusion of paracetamol or placebo. | up to 4 hours

SECONDARY OUTCOMES:
Assessment of time interval of pain < 4 on the NRS (after been achieved) | up to 4 hours
Total dose of morphine within the first 4 hours after the first infusion of paracetamol or Placebo. | up to 4 hours
Prevalence of morphine adverse reactions within the first 4 hours after infusion of paracetamol or placebo | up to 4 hours, respectively in case of serious adverse events up to recovery time of the patient

OTHER OUTCOMES:
Maximal Dose of Morphine based on adverse events | up to 4 hours
  A maximal Dose of opioids has been defined in our daily practice and in several guidelines with a precise number (e.g. 20 mg/4 h). In this trial we will use instead a maximal Dose defined with clinical criteria (GCS < 13, SpO2 < 90% with 4 L/min O2, uncontrolled vomiting). Assessment intended as occurrence of adverse events of the application of a such algorithms will be outcome of interest (not a secondary outcome because absence of a control group)

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No